CLINICAL TRIAL: NCT01437202
Title: Retrospective Study to Validate Pharmacogenetics Model for Imatinib Metabolism in Patients With Chronic Myeloid Leukemia
Brief Title: Pharmacogenomics Validation for Imatinib in Chronic Myeloid Leukemia
Acronym: VATIC
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Dae-Young Kim, Assistant Professor, Asan Medical Center
Other Study IDs: AMC-H-64
Record Dates: First submitted 2011-09-19; First posted 2011-09-20 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Leukemia, Myelogenous, Chronic, BCR-ABL Positive
Keywords: imatinib; drug resistance; pharmacogenetics
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood 4cc
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- high risk group: Identified by the predictive model using 2 genotypes and disease stage
- intermediate risk group: Identified by the predictive model using 2 genotypes and disease stage
- Low risk group: Identified by the predictive model using 2 genotypes and disease stage

SUMMARY:
This is a multicenter, retrospective, observational study to validate a pharmacogenetics model for imatinib metabolism and resistance in patients with chronic myeloid leukemia among patients in different independent cohort.

DETAILED DESCRIPTION:
1. The activity of Imatinib(IM) is mediated by blocking the activity of BCR/ABL tyrosine kinase in CML cells. However, some of the patients failed to achieve optimal response, and a substantial proportion of patients develop resistance to IM.
2. IM is a substrate for the adenosine triphosphate binding cassette (ABC) transporters, ABCB1 and ABCG2, while the active uptake of IM into cells is mediated by the human organic cationic transporter-1 (hOCT1). Also, IM is metabolized through first pass drug metabolism by the cytochrome P450 - CYP3A4 and CYP3A5. In addition, it is delivered in a bound form with a plasma protein referred to α1-acid glycoprotein (AGP).
3. Accordingly, the intracellular or systemic level of imatinib should be influenced by these factors such as ABCB1, ABCG2, hOCT1, CYP3A4, CYP3A5 or AGP genes. Inter-individual variability of 5 candidate genes associated with drug transport/metabolism (i.e. ABCB1, ABCG2, hOCT1, CYP3A4/3A5 and AGP) could affect the expression of corresponding proteins, thus influencing the treatment outcomes of imatinib therapy.
4. In the investigators' previous study, the investigators reported the cumulative incidences of MCyR and CCyR was significantly affected by the predictive model using 2 genotypes and disease stage. These predictive models for CCyR/MMoR or LOR/treatment failure seemed to work well. However, external validation of these predictive models is warranted especially using ethnically different independent cohort.

ELIGIBILITY:
Inclusion Criteria:

* Chronic myeloid leukemia of any stage including chronic phase, accelerated or blastic phase.
* Age>18 years
* Complete set of clinical data available for review (demographic data, stage, treatment history, cytogenetic reports, and latest BCR/ABL RQ-PCR results)
* Treated with imatinib mesylate at least 3 months

Exclusion Criteria:

* Treated with imatinib mesylate less than 3 months
* Not agree with the intention of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed as chronic myeloid leukemia, treated with imatinib more than 3 months, at Asan Medical Center, Seoul, Korea.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Median time to CCyR (complete cytogenetic response)
  Difference of median time to CCyR between cohorts according to the risk stratification by gene analysis

SECONDARY OUTCOMES:
Variance of Genotypes from CML patients with Korean ethnicity
Median time to MCyR (Major cytogenetic responses)
  Difference of median time to MCyR between cohorts according to the risk stratification by gene analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jong Won Kim, MD, PhD, Study Chair — Samsung Medical Center, Sungjyunkwan University School of Medicine, Seoul, Korea; Dae-Young Kim, MD, Principal Investigator — Asan Medical Center, University of Ulsan College of Medicine, Seoul, Korea
Locations (3):
- Princess Margaret Hospital, University of Toronto, Toronto, Canada
- South Korea (2):
  - Asan Medical Center, University of Ulsan College of Medicine, Seoul
  - Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul

REFERENCES:
- [Background] Kantarjian HM, Cortes JE, O'Brien S, Luthra R, Giles F, Verstovsek S, Faderl S, Thomas D, Garcia-Manero G, Rios MB, Shan J, Jones D, Talpaz M. Long-term survival benefit and improved complete cytogenetic and molecular response rates with imatinib mesylate in Philadelphia chromosome-positive chronic-phase chronic myeloid leukemia after failure of interferon-alpha. Blood. 2004 Oct 1;104(7):1979-88. doi: 10.1182/blood-2004-02-0711. Epub 2004 Jun 15. PMID 15198956
- [Background] Kantarjian HM, Talpaz M, Giles F, O'Brien S, Cortes J. New insights into the pathophysiology of chronic myeloid leukemia and imatinib resistance. Ann Intern Med. 2006 Dec 19;145(12):913-23. doi: 10.7326/0003-4819-145-12-200612190-00008. PMID 17179059
- [Background] Gorre ME, Mohammed M, Ellwood K, Hsu N, Paquette R, Rao PN, Sawyers CL. Clinical resistance to STI-571 cancer therapy caused by BCR-ABL gene mutation or amplification. Science. 2001 Aug 3;293(5531):876-80. doi: 10.1126/science.1062538. Epub 2001 Jun 21. PMID 11423618
- [Background] Mahon FX, Belloc F, Lagarde V, Chollet C, Moreau-Gaudry F, Reiffers J, Goldman JM, Melo JV. MDR1 gene overexpression confers resistance to imatinib mesylate in leukemia cell line models. Blood. 2003 Mar 15;101(6):2368-73. doi: 10.1182/blood.V101.6.2368. PMID 12609962
- [Background] Awidi A, Salem II, Najib N, Mefleh R, Tarawneh B. Determination of imatinib plasma levels in patients with chronic myeloid leukemia by high performance liquid chromatography-ultraviolet detection and liquid chromatography-tandem mass spectrometry: methods' comparison. Leuk Res. 2010 Jun;34(6):714-7. doi: 10.1016/j.leukres.2009.08.005. Epub 2009 Sep 9. PMID 19744707
- [Background] Gardner ER, Burger H, van Schaik RH, van Oosterom AT, de Bruijn EA, Guetens G, Prenen H, de Jong FA, Baker SD, Bates SE, Figg WD, Verweij J, Sparreboom A, Nooter K. Association of enzyme and transporter genotypes with the pharmacokinetics of imatinib. Clin Pharmacol Ther. 2006 Aug;80(2):192-201. doi: 10.1016/j.clpt.2006.05.003. PMID 16890580
- [Result] Kim DH, Sriharsha L, Xu W, Kamel-Reid S, Liu X, Siminovitch K, Messner HA, Lipton JH. Clinical relevance of a pharmacogenetic approach using multiple candidate genes to predict response and resistance to imatinib therapy in chronic myeloid leukemia. Clin Cancer Res. 2009 Jul 15;15(14):4750-8. doi: 10.1158/1078-0432.CCR-09-0145. Epub 2009 Jul 7. PMID 19584153